**Statistical Analysis Plan** 

Title: Analgesic Effects of Intranasal Diclofenac Sodium, Ibuprofen, and Paracetamol in Pediatric

**Tonsillectomy Cases** 

Document Date: 11/12/2024

NCT Number: NCT06731556

Unique Protocol ID: 20.08.2021-E.28962

Objectives:

-Assess the efficacy of intranasal NSAIDs compared to intravenous paracetamol.

-Evaluate safety and side effects.

Population:

-60 pediatric patients divided into four groups.

Statistical Methods:

Descriptive statistics of the quantitative variables in the study are presented as mean, median,

standard deviation, minimum, and maximum. The compatibility of the variables with normal

distribution was analyzed using the Kolmogorov-Smirnov test. The Kruskal-Wallis test was

employed to compare the means of the related variables between independent groups containing

more than two groups. Dunn's test was used as a post hoc analysis for multiple comparisons.

Similarly, the Kruskal-Wallis and Dunn's tests were utilized for group comparisons in terms of

mean changes between periods. The statistical significance level was set at 0.05, and IBM SPSS

(version 26) software was used for all calculations. A p-value of less than 0.05 was considered

statistically significant.

Handling Missing Data:

- Missing values to be handled by exclusion from specific analyses.